CLINICAL TRIAL: NCT01562769
Title: Interest of Contact Precautions for Preventing Micro-organisms Acquisition in Patients Hospitalized in Infectious Disease Unit of University-affiliated Hospital in Rennes
Acronym: ISOL/STAND
Status: Terminated | Type: Observational
Why Stopped: enrollment difficulties
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-A01360-41; LOC/11-20 (Other: Rennes University Hospital (Direction of Clinical Research))
Record Dates: First submitted 2012-03-22; First posted 2012-03-26 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-05

CONDITIONS: Patients Hospitalized in Infectious Disease

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Standard precautions: One selected part of the unit keep the usual procedure applied in our institution with contact precautions prescriptions when colonized patient is admitted with SA and/or ESBL bacteria.
  Second selected part of the unit applies only standard precautions (even for patients colonized with multiple drug-resistant organisms).
  After 8 months precaution procedures will be exchanged between the two sectors (cross over design).
- contact precautions: One selected part of the unit keep the usual procedure applied in our institution with contact precautions prescriptions when colonized patient is admitted with SA and/or ESBL bacteria.
  Second selected part of the unit applies only standard precautions (even for patients colonized with multiple drug-resistant organisms).
  After 8 months precaution procedures will be exchanged between the two sectors (cross over design).

SUMMARY:
Application of isolation (=contact precautions) in hospitalized patients is recommended when patient is colonized (or infected) by micro-organism known for its outbreak capacity or high pathogenicity. It allows the reinforcement of universal precautions (=standard precautions) in order to control patient-to-patient micro-organisms transmission. Recently, the efficacy of this measure is questioned and its impact on patient care seems deleterious.

In a particular context of Infectious Disease Unit, where standard precautions are handled (favorable architecture and appropriate practice for hand hygiene), assessment of contact precautions to reduce the incidence of acquired bacteria during hospitalization would be of interest.

The investigators design a non-inferiority comparative study to measure the colonization pressure in patients hospitalized in two different parts of the department: one unit only with standard precautions applied (intervention) and one unit with contact precautions (control) as current routine care.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized in Infectious Diseases Unit during the study period in one of the selected part of the unit participating to the study
* Patient informed about the study protocol and approved to participate.

Exclusion Criteria:

* Patient requiring isolation prescription type "air" or "droplet"
* Patient hospitalized in the central sector of the building (including 4 bedrooms in depression negative service)
* Patient colonized with bacteria producing carbapenemase, multi-resistant Acinetobacter baumanii or Vancomycin-Resistant Enterococcus.
* Patients under legal protection (juridical protection, legal guardianship) or persons on juridical detention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in Infectious Disease Unit of university-affiliated hospital in Rennes
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2012-03; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Acquisition rate of micro-organisms | 2 years
  Acquisition rate using bacteriological sampling (nose and anus) at admission and at the day of discharge in each patient hospitalized in the department.

SECONDARY OUTCOMES:
Number of infections acquired during hospitalization in each group | 2 years
Consumption of hydro-alcoholic rub in each group | 2 years
Utilization of aprons and gloves in each group | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: jean-marc chapplain, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, Brittany Region, France